CLINICAL TRIAL: NCT02920034
Title: A Randomized Comparison of Ultrasound Based Versus Radiofrequency Based Catheter Ablation Techniques in Patients With Therapy Resistant Arterial Hypertension With Large Renal Arteries
Brief Title: Randomized Comparison of Ultrasound Versus Radiofrequency Denervation in Patients With Therapy Resistant Hypertension
Acronym: RADIOSOUND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Philipp Lurz, Clinical Investigator, Professor, Managing Senior Physician, Heart Center Leipzig - University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Radiosound 1.1
Record Dates: First submitted 2016-09-24; First posted 2016-09-30 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Therapy Resistant Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Radiofrequency main renal artery (Active Comparator): Renal sympathetic denervation of the main renal artery using the radiofrequency-based Spyral™ catheter (Medtronic, MN, USA)
  Interventions: Device: Radiofrequency denervation of the main renal arteries
- Radiofrequency main and branches (Experimental): Renal sympathetic denervation of the main renal artery, its branches and accessories using the radiofrequency-based Spyral™ catheter (Medtronic, MN, USA)
  Interventions: Device: Radiofrequency denervation of renal arteries and branches
- Ultrasound main renal artery (Experimental): Renal sympathetic denervation of the main renal artery using the ultrasound-based Paradise™ catheter (ReCor, CA, USA)
  Interventions: Device: Ultrasound denervation of the main renal arteries

INTERVENTIONS:
Device: Radiofrequency denervation of the main renal arteries — Catheter based renal sympathetic denervation of the main renal arteries using the Spyral™ Catheter (Medtronic, MN, USA)
  Arms: Radiofrequency main renal artery
Device: Radiofrequency denervation of renal arteries and branches — Catheter based renal sympathetic denervation of the main renal arteries and its branches using the Spyral™ Catheter (Medtronic, MN, USA)
  Arms: Radiofrequency main and branches
Device: Ultrasound denervation of the main renal arteries — Catheter based renal sympathetic denervation of the main renal arteries using the Paradise™ Catheter (ReCor Medical, CA, USA)
  Arms: Ultrasound main renal artery

SUMMARY:
Prospective, randomized trial to assess the effectiveness of different renal sympathetic denervation methods (radiofrequency main vs. branches + main vs. ultrasound based) in a cohort of patients with therapy refractory arterial hypertension and large renal arteries

DETAILED DESCRIPTION:
The aim of this trial is a prospective, randomized comparison of three different techniques for catheter based renal sympathetic denervation. Patients with larger (>5.5 mm) renal arteries are randomized to a treatment with a radiofrequency based catheter of the main renal artery, the main renal artery, its side-branches and accessories or an ultrasound-based denervation of the main renal artery only. The primary endpoint is the change in daytime blood pressure acquired in ambulatory blood pressure measurement at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resistant hypertension (≥3 antihypertensive drugs including at least one diuretic, without any dosage change in the preceding 4 weeks) and a systolic office blood pressure of >160 mmHg, ≥1 main renal artery diameter >5.5 mm

Exclusion Criteria:

* pregnancy, known renal artery stenosis, average systolic daytime RR <135 mmHg in 24h ambulatory blood pressure measurement (ABPM), ≥1 renal artery diameter <4.0 mm, life-expectancy <6 months, participation in any other clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Daytime blood pressure change | 3 months after Intervention
  Daytime blood pressure change in ambulatory blood pressure measurement

SECONDARY OUTCOMES:
General blood pressure change | 3 months after Intervention
  Change in 24 h average blood pressure change in ambulatory blood pressure measurement
Daytime blood pressure change | 6 months after Intervention
  Daytime blood pressure change in ambulatory blood pressure measurement
General blood pressure change | 6 months after Intervention
  Change in 24 h average blood pressure change in ambulatory blood pressure measurement
Daytime blood pressure change | 12 months after Intervention
  Daytime blood pressure change in ambulatory blood pressure measurement
Daytime blood pressure change | 24 months after Intervention
  Daytime blood pressure change in ambulatory blood pressure measurement
General blood pressure change | 12 months after Intervention
  Change in 24 h average blood pressure change in ambulatory blood pressure measurement
General blood pressure change | 24 months after Intervention
  Change in 24 h average blood pressure change in ambulatory blood pressure measurement
Exercise blood pressure change | 3 months after Intervention
  Change in exercise blood pressure on bicycle stress testing

CONTACTS AND LOCATIONS:
Overall Officials: Philipp C Lurz, MD, PhD, Principal Investigator — Heart Center of the University Leipzig
Locations (1):
- Heart Center of the University Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fengler K, Rommel KP, Kriese W, Blazek S, Besler C, von Roeder M, Desch S, Thiele H, Lurz P. 6- and 12-Month Follow-Up From a Randomized Clinical Trial of Ultrasound vs Radiofrequency Renal Denervation (RADIOSOUND-HTN). JACC Cardiovasc Interv. 2023 Feb 13;16(3):367-369. doi: 10.1016/j.jcin.2022.10.058. No abstract available. PMID 36792266
- [Derived] Fengler K, Rommel KP, Lapusca R, Blazek S, Besler C, Hartung P, von Roeder M, Kresoja KP, Desch S, Thiele H, Lurz P. Renal Denervation in Isolated Systolic Hypertension Using Different Catheter Techniques and Technologies. Hypertension. 2019 Aug;74(2):341-348. doi: 10.1161/HYPERTENSIONAHA.119.13019. Epub 2019 Jun 17. PMID 31203726
- [Derived] Fengler K, Rommel KP, Blazek S, Besler C, Hartung P, von Roeder M, Petzold M, Winkler S, Hollriegel R, Desch S, Thiele H, Lurz P. A Three-Arm Randomized Trial of Different Renal Denervation Devices and Techniques in Patients With Resistant Hypertension (RADIOSOUND-HTN). Circulation. 2019 Jan 29;139(5):590-600. doi: 10.1161/CIRCULATIONAHA.118.037654. PMID 30586691